CLINICAL TRIAL: NCT02505555
Title: Accuracy and Tolerability of Four-dimensional Hysterosalpingo-contrast Sonography With SonoVue for Assessment of Tubal Patency
Brief Title: Feasibility of Four-dimensional Hysterosalpingo-contrast Sonography With SonoVue for Assessment of Tubal Patency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Bai Wen-Pei, Professor,Chief of Obstetrics and Gynecology Department, Peking University First Hospital
Other Study IDs: PekingUFH-4DF; 4D-HyCoSy (Other: PekingUFH)
Record Dates: First submitted 2015-07-04; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Four Dimensional Hysterosalpingo-contrast Sonography; Tubal Patency
Keywords: feasibility; accuracy; tolerability; four dimensional hysterosalpingo-contrast sonography

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: four dimensional hysterosalpingo-contrast sonography — compare accuracy and tolerability of 4D-HyCoSy with that of laparoscopy and chromotubation
  Other Names: 4D-HyCoSy

SUMMARY:
The purpose of this study is to summarize our experience with and to evaluate the feasibility of transvaginal four-dimensional hysterosalpingo-contrast sonography using SonoVue (4D-HyCoSy) for assessment of fallopian tubal patency, women attending the fertility clinic are recruited. All of the patients are tried to be examined with 4D-HyCoSy,some of who undergone laparoscopy and dye. Then the results of 4D-HyCoSy and lap and dye are compared. All of the patients will be followed up. The complications of 4D-HyCoSy will be evaluated and the pregnancy outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women who have infertility and need to evaluate tubal patency.

Exclusion Criteria:

1. vaginal bleeding;
2. acute or subacute inflammation of the reproductive system;
3. uterine malignancies;
4. allergies to the medications used in the examination, such as lidocaine, atropine, and sulfur hexafluoride

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who have infertility and try to evaluate tubal patency by 4D-HyCoSy in our hospital will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of four-dimensional hysterosalpingo-contrast sonography with SonoVue | at least one year
  Sensitivity, specificity, accuracy, positive predictive value, negative predictive value

SECONDARY OUTCOMES:
side effects and complications of four-dimensional hysterosalpingo-contrast sonography | at least one year
  the intensity of pain perception, vaginal bleeding, fever, pelvic inflammatory diseases，peritonitis，and the pregnancy outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Marana R, Ferrari S, Merola A, Astorri AL, Pompa G, Milardi D, Giampietro A, Lecca A, Marana E. [Role of a mini-invasive approach in the diagnosis and treatment of tubo-peritoneal infertility as an altenative to IVF]. Minerva Ginecol. 2011 Feb;63(1):1-10. Italian. PMID 21311415
- [Result] Luciano DE, Exacoustos C, Luciano AA. Contrast ultrasonography for tubal patency. J Minim Invasive Gynecol. 2014 Nov-Dec;21(6):994-8. doi: 10.1016/j.jmig.2014.05.017. Epub 2014 Jun 6. PMID 24910933
- [Result] Maheux-Lacroix S, Boutin A, Moore L, Bergeron ME, Bujold E, Laberge P, Lemyre M, Dodin S. Hysterosalpingosonography for diagnosing tubal occlusion in subfertile women: a systematic review with meta-analysis. Hum Reprod. 2014 May;29(5):953-63. doi: 10.1093/humrep/deu024. Epub 2014 Feb 26. PMID 24578476
- [Result] Exacoustos C, Di Giovanni A, Szabolcs B, Romeo V, Romanini ME, Luciano D, Zupi E, Arduini D. Automated three-dimensional coded contrast imaging hysterosalpingo-contrast sonography: feasibility in office tubal patency testing. Ultrasound Obstet Gynecol. 2013 Mar;41(3):328-35. doi: 10.1002/uog.11200. PMID 22648792
- [Result] He Y, Geng Q, Liu H, Han X. First experience using 4-dimensional hysterosalpingo-contrast sonography with SonoVue for assessing fallopian tube patency. J Ultrasound Med. 2013 Jul;32(7):1233-43. doi: 10.7863/ultra.32.7.1233. PMID 23804346
- [Result] Tur-Kaspa I. Fear no pain: uterine cavity and tubal patency assessment tests should be pain free. Ultrasound Obstet Gynecol. 2012 Mar;39(3):247-51. doi: 10.1002/uog.11128. No abstract available. PMID 22535627
- [Result] Marci R, Marcucci I, Marcucci AA, Pacini N, Salacone P, Sebastianelli A, Caponecchia L, Lo Monte G, Rago R. Hysterosalpingocontrast sonography (HyCoSy): evaluation of the pain perception, side effects and complications. BMC Med Imaging. 2013 Aug 23;13:28. doi: 10.1186/1471-2342-13-28. PMID 23968513
- [Result] Socolov D, Boian I, Boiculese L, Tamba B, Anghelache-Lupascu I, Socolov R. Comparison of the pain experienced by infertile women undergoing hysterosalpingo contrast sonography or radiographic hysterosalpingography. Int J Gynaecol Obstet. 2010 Dec;111(3):256-9. doi: 10.1016/j.ijgo.2010.07.018. Epub 2010 Sep 17. PMID 20850745
- [Result] Giugliano E, Cagnazzo E, Bazzan E, Patella A, Marci R. Hysterosalpingo-contrast sonography: is possible to quantify the therapeutic effect of a diagnostic test? Clin Exp Reprod Med. 2012 Dec;39(4):161-5. doi: 10.5653/cerm.2012.39.4.161. Epub 2012 Dec 31. PMID 23346526
- [Result] O'Flynn N. Assessment and treatment for people with fertility problems: NICE guideline. Br J Gen Pract. 2014 Jan;64(618):50-1. doi: 10.3399/bjgp14X676609. No abstract available. PMID 24567574
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Marana%2C+R.%2C+et+al.%2C+%5BRole+of+a+mini-invasive+approach+in+the+diagnosis+and+treatment+of+tubo-peritoneal+infertility+as+an+altenative+to+IVF%5D.+Minerva+Ginecol%2C+2011.+63(1)%3A+p.+1-10.